CLINICAL TRIAL: NCT02832986
Title: Herpes Zoster Prevalence in Frailty Consultations in University Hospital of Toulouse
Brief Title: Herpes Zoster Prevalence in Frailty Consultations
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31-15-7581
Record Dates: First submitted 2016-07-01; First posted 2016-07-14 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Herpes Zoster
Keywords: Frailty consultation
MeSH Terms: conditions — Herpes Zoster

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients in frailty consultation: Patients consulting in frailty consultation, at this occasion they will complete a medical questionary for the collection of study data
  Interventions: Other: Medical Questionary

INTERVENTIONS:
Other: Medical Questionary — The medical questionary will contain :
  * Date of initial infection by Herpes zoster
  * Localisation
  * Severity
  * Presence of postherpetic pain
  * Postherpetic pain Intensity
  * Postherpetic pain duration
  * Antiviral treatment
  * History of chronic pathologies
  * Concomitant treatment

SUMMARY:
Herpes zoster and post herpetic pain are common causes of morbidity in the elderly. Herpes zoster is caused by reactivation of the virus varicella zoster of latent infection in sensory ganglia. The acute phase of herpes zoster usually occurs ≤ 30 days after rash onset. However, the most common complication of herpes zoster is the post herpetic pain, which is usually defined as a persistent chronic pain for ≥ 3 months after rash onset. The risk of herpes zoster in life is 25-30%, but this figure rises to 50% among those aged ≥ 85 years. Similarly, the risk of experiencing post herpetic pain increases with age.

Despite treatment with antiviral drugs, post herpetic pain has been reported in 10-20% of all patients with herpes zoster, but its incidence increases significantly in elderly patients over 60 years. It can be particularly harmful when it occurs on a particular field, elderly multiple pathologies, fragile and with multiple treatment. In this context of decompensation "cascade" greatly exacerbate the impact of the initial local disease. Ophthalmologic involvement is rare but clinically worrisome and generates significant costs.

DETAILED DESCRIPTION:
The annual incidence of herpes zoster in France is estimated at 3.4-4.4 cases per 1 000 people in the general population regardless of the history of Herpes zoster. The highest incidence concerns people aged 65 and over with an incidence estimated between 8-10 cases per 1 000 people, representing more than 100 000 cases of herpes zoster.

Due to the increasing number of older people in the French population, the number of herpes zoster should thus parallel increase in the coming years. The risk factors are well identified for certain (age, ethnicity ...) but for others less well defined (diabetes, composite criteria multiple pathologies ...) and insufficient to explain why some people exposed to the same risk factors will not make shingles during their lifetime.

Post herpetic pain is the leading complication of this disease with a higher risk in patients over 70 years causing a risk of autonomy loss. In fact, besides the disability of the pain itself, post herpetic pain often requires a combination of high-dose painkillers. The main therapeutic classes of analgesics used are antiepileptic in high doses (Gabapentin, Pregabalin), tricyclic antidepressants (amitriptyline), or opiates. The prevention with herpes zoster vaccine showed a reduction by 2 of risk and could therefore prevent addiction caused by induced recurrences of herpes zoster and treatment of post herpetic pain.

A study of importance is needed to further define the prevalence of this disease in the population of frail elderly and to identify factors associated with the occurrence of herpes zoster, post herpetic pain and ophthalmic zoster.

ELIGIBILITY:
Inclusion Criteria:

* Patients consulting at the daily hospital of fragility and dependence prevention during inclusion period

Exclusion Criteria:

* Patients not consulting daily hospital of fragility and dependence prevention
* Patients consulting outside the inclusion period dates
* Patients vaccinated against zoster

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients consulting in frailty consultation
Sampling Method: Non-Probability Sample
Enrollment: 1245 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Frequence of zoster antecedent as assessed by percentage of subject with zoster antecedent | Day 1
  During the frailty consultation

SECONDARY OUTCOMES:
Frequence of ophthalmic zoster antecedent as assessed by percentage of subject with ophthalmic zoster antecedent | Day 1
  During the frailty consultation
Frequence of postherpetic pain antecedent as assessed by percentage of subject with postherpetic pain antecedent | Day 1
  During the frailty consultation
Risk factor associated with herpes zoster antecedent by usage of logistic regression model | Through the completion of study (12 months)
  Proportion of herpes zoster antecedents and characteristics will be defined by percentage of patient with medical data confirming antecedents of herpes zoster
Risk factor associated with postherpetic pain by usage of logistic regression model | Through the completion of study (12 months)
Risk factor associated with ophthalmic zoster by usage of logistic regression model | Through the completion of study (12 months)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno VELLAS, MD, Principal Investigator — University Hospital of Toulouse
Locations (1):
- University Hospital of Toulouse - geriatric pole, Toulouse, France

IPD SHARING:
Plan to Share IPD: Undecided